CLINICAL TRIAL: NCT00779103
Title: Phase III, Open-Label Study to Evaluate Efficacy and Safety of Histrelin Subdermal Implant in Children With Central Precocious Puberty
Brief Title: Histrelin Subcutaneous Implant in Children With Central Precocious Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3326-300Former03-CPP-HIS-300
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-10

CONDITIONS: Central Precocious Puberty
Keywords: puberty; precocious puberty; early puberty; early onset puberty; histrelin; histrelin subcutaneous implant; implant therapy
MeSH Terms: conditions — Puberty, Precocious | interventions — histrelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Histrelin Subcutaneous Implant (50 mg) (Experimental): Subcutaneous implant designed to deliver histrelin continously for 12 months.
  Interventions: Drug: Histrelin Subcutaneous Implant

INTERVENTIONS:
Drug: Histrelin Subcutaneous Implant — histrelin subcutaneous 50 mg implant
  Other Names: Supprelin LA; implant therapy; histrelin implant

SUMMARY:
The purpose of this study is to follow and collect additional medical and developmental information on children after histrelin subcutaneous implant therapy is discontinued.

DETAILED DESCRIPTION:
Thirty-two (32) patients will receive a histrelin subdermal implant under the anesthesia deemed appropriate by the administering physician. Ten-twelve (10-12) sites will enroll 2-3 patients per site. It is anticipated that half the patients will be receiving GnRH analog treatment and the other half will be treatment naïve. All patients will undergo selective PK sampling post-implantation to assess histrelin profile. At 12 months, provided that the patient continues to meet the safety and efficacy parameters, the original implant will be removed and the patient can receive a new implant. At 13 months, patients who receive new implants will be evaluated at the study site and administratively transferred to the initial extension study. At Month 24), the implants inserted at Month 12 will be removed. At this time, patients who have completed the initial extension study and who wish to continue therapy with the histrelin implant will be eligible to receive a new (ie, third) implant and to enter an additional 12-month extended access phase at the discretion of the investigator. At Month 36, the implants inserted at Month 24 for the Extended Access Phase will be removed. At this time, patients who have completed the Extended Access Phase and who wish to continue therapy with the histrelin implant will be eligible to receive a new (ie, fourth) implant and to enter the Long Term Extended Access Phase (referred to as the Implant Treatment Phase) at the discretion of the investigator. The purpose of this phase is to provide patients with the opportunity to continue to receive a new implant at the end of each 12-month period until the patient no longer requires hormone suppression. Once implant therapy is discontinued, all patients are eligible to enter the Long Term Follow Up Phase (Post Implant Phase) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre-treated or treatment naive patients with gonadotropin-dependent precocious puberty
* Pre-treatment pubertal type response of LH to a stndard GnRH stimulation test before initiation of treatment

Exclusion Criteria:

* Children who are less than 2 years of age at enrollment
* Children whose chronological age is greater than 8 years (naive) and 10 years (pre-treated) for girls or 9 years (naive) and 11 years (pre-treated) for boys at the onset of the study

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2004-09; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica A Eugster, MD, Principal Investigator — Indiana University School of Medicine, 705 Riley Hosp Dr, Rm 5960 Indianapolis, IN 46202

REFERENCES:
- [Derived] Silverman LA, Neely EK, Kletter GB, Lewis K, Chitra S, Terleckyj O, Eugster EA. Long-Term Continuous Suppression With Once-Yearly Histrelin Subcutaneous Implants for the Treatment of Central Precocious Puberty: A Final Report of a Phase 3 Multicenter Trial. J Clin Endocrinol Metab. 2015 Jun;100(6):2354-63. doi: 10.1210/jc.2014-3031. Epub 2015 Mar 24. PMID 25803268
- [Derived] Neely EK, Silverman LA, Geffner ME, Danoff TM, Gould E, Thornton PS. Random unstimulated pediatric luteinizing hormone levels are not reliable in the assessment of pubertal suppression during histrelin implant therapy. Int J Pediatr Endocrinol. 2013 Dec 2;2013(1):20. doi: 10.1186/1687-9856-2013-20. PMID 24295437

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall - Histrelin Subcutaneous Implant (50 mg): Subcutaneous implant designed to deliver histrelin continously for 12 months.
  Histrelin Subcutaneous Implant: histrelin subcutaneous 50 mg implant
Period: Overall Study
Arm/Group | Overall - Histrelin Subcutaneous Implant (50 mg)
Started | 36 (Initial Phase (First Implant) - 36 Completed)
Second & Third Implant | 31 (Initial Extension Phase/Extended Access Phase (Second and Third Implant) - 22 Completed)
Fourth Implant | 13 (Second Extension Phase (4th Implant with Yearly Implantations till no longer required): 11 Completed)
No Treatment | 9 (Optional Long Term Follow-up Phase (No Treatment))
Completed | 36 (Initial Phase (First Implant))
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Initial Extension Phase/Extended Access Phase (Second and Third Implant)
Groups:
- Histrelin Subcutaneous Implant (50 mg): Subcutaneous implant designed to deliver histrelin continously for 12 months.
  Histrelin Subcutaneous Implant: histrelin subcutaneous 50 mg implant
  Extension Safety Population (Second & Third Implant)
Arm/Group | Histrelin Subcutaneous Implant (50 mg)
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 1
  Unknown or Not Reported | 13
Height [Mean (Standard Deviation); unit: cm] | 134.18 (12.947)
Weight [Mean (Standard Deviation); unit: kg] | 38.12 (11.835)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 20.66 (3.541)
Pretreatment with Prior GnRH Therapy [Count of Participants; unit: Participants]
  Pretreated | 13
  Naïve | 18

OUTCOME MEASURES:

1. Primary Outcome: Luteinizing Hormone (LH)
Description: The suppression of gonadotropins (luteinizing hormone and follicle stimulating hormone) and gonadal sex steroids (estrogen in girls and testosterone in boys, respectively) on treatment.(LH suppression is defined as a peak LH < 4 mIU/mL following stimulation with the GnRH analog).
Time Frame: Baseline - 6 Months Post Last Implant
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: MIU/ML
Arm/Group | Observed Value | Change From Baseline
Number analyzed (Participants) | 31 | 31
MIU/ML
  Baseline: number analyzed (Participants) | 31 | 0
  Baseline | 0.88 (1.244) |
  Day 1, Visit 1: number analyzed (Participants) | 1 | 1
  Day 1, Visit 1 | 0.53 | 0.07
  Month 1, Visit 2 | 0.50 (0.302) | -0.37 (1.111)
  Month 3, Visit 3: number analyzed (Participants) | 30 | 30
  Month 3, Visit 3 | 0.39 (0.247) | -0.50 (1.173)
  Month 6, Visit 4: number analyzed (Participants) | 30 | 30
  Month 6, Visit 4 | 0.37 (0.225) | -0.53 (1.227)
  Month 9, Visit 5: number analyzed (Participants) | 30 | 30
  Month 9, Visit 5 | 0.38 (0.266) | -0.51 (1.170)
  Month 12, Visit 6 | 0.38 (0.247) | -0.50 (1.108)
  Month 13, Visit 7: number analyzed (Participants) | 29 | 29
  Month 13, Visit 7 | 0.35 (0.216) | -0.58 (1.217)
  Month 18, Visit 9: number analyzed (Participants) | 29 | 29
  Month 18, Visit 9 | 0.24 (0.118) | -0.68 (1.233)
  Month 24, Visit 11 | 0.22 (0.124) | -0.66 (1.228)
  Month 36, Visit 13: number analyzed (Participants) | 13 | 13
  Month 36, Visit 13 | 0.19 (0.126) | -0.42 (0.734)
  Month 42, Visit 14: number analyzed (Participants) | 10 | 10
  Month 42, Visit 14 | 0.14 (0.119) | -0.53 (0.842)
  Month 48, Visit 15: number analyzed (Participants) | 12 | 12
  Month 48, Visit 15 | 0.25 (0.232) | -0.36 (0.871)
  Month 54, Visit 16: number analyzed (Participants) | 4 | 4
  Month 54, Visit 16 | 0.24 (0.272) | -0.47 (1.402)
  Month 60, Visit 17: number analyzed (Participants) | 9 | 9
  Month 60, Visit 17 | 0.27 (0.336) | -0.24 (0.937)
  Month 66, Visit 18: number analyzed (Participants) | 2 | 2
  Month 66, Visit 18 | 0.18 (0.020) | 0.07 (0.100)
  Month 72, Visit 19: number analyzed (Participants) | 2 | 2
  Month 72, Visit 19 | 0.36 (0.357) | 0.26 (0.237)
  1 Month Post Last Implant: number analyzed (Participants) | 8 | 8
  1 Month Post Last Implant | 0.81 (0.952) | 0.53 (0.958)
  6 Month Post Last Implant: number analyzed (Participants) | 8 | 8
  6 Month Post Last Implant | 3.66 (2.463) | 3.38 (2.410)

2. Secondary Outcome: Follicle Stimulating Hormone (FSH)
Description: as for outcome 1
Time Frame: Baseline - 6 Month Post Last Implant
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: MIU/ML
Arm/Group | Observed Value | Change From Baseline
Number analyzed (Participants) | 31 | 31
MIU/ML
  Baseline: number analyzed (Participants) | 31 | 0
  Baseline | 2.26 (1.656) |
  Day 1, Visit 1: number analyzed (Participants) | 1 | 1
  Day 1, Visit 1 | 1.60 | -0.20
  Month 1, Visit 2 | 1.08 (0.611) | -1.18 (1.566)
  Month 3, Visit 3 | 1.36 (0.814) | -0.90 (1.464)
  Month 6, Visit 4: number analyzed (Participants) | 30 | 30
  Month 6, Visit 4 | 1.43 (0.787) | -0.86 (1.674)
  Month 9, Visit 5: number analyzed (Participants) | 30 | 30
  Month 9, Visit 5 | 1.77 (0.939) | -0.52 (1.776)
  Month 12, Visit 6 | 2.16 (1.712) | -0.10 (1.868)
  Month 13, Visit 7: number analyzed (Participants) | 29 | 29
  Month 13, Visit 7 | 1.68 (1.048) | -0.65 (1.394)
  Month 18, Visit 9: number analyzed (Participants) | 29 | 29
  Month 18, Visit 9 | 1.81 (1.142) | -0.50 (1.668)
  Month 24, Visit 11 | 1.89 (0.855) | -0.37 (1.486)
  Month 36, Visit 13: number analyzed (Participants) | 14 | 14
  Month 36, Visit 13 | 1.91 (1.146) | -0.01 (1.027)
  Month 42, Visit 14: number analyzed (Participants) | 10 | 10
  Month 42, Visit 14 | 1.63 (1.119) | -0.62 (1.457)
  Month 48, Visit 15: number analyzed (Participants) | 12 | 12
  Month 48, Visit 15 | 1.55 (1.199) | -0.48 (1.619)
  Month 54, Visit 16: number analyzed (Participants) | 5 | 5
  Month 54, Visit 16 | 1.43 (0.752) | -0.73 (2.288)
  Month 60, Visit 17: number analyzed (Participants) | 9 | 9
  Month 60, Visit 17 | 1.50 (0.741) | -0.57 (1.573)
  Month 66, Visit 18: number analyzed (Participants) | 2 | 2
  Month 66, Visit 18 | 0.76 (0.049) | -0.89 (1.578)
  Month 72, Visit 19: number analyzed (Participants) | 2 | 2
  Month 72, Visit 19 | 1.24 (0.369) | -0.41 (1.257)
  1 Month Post Last Implant: number analyzed (Participants) | 8 | 8
  1 Month Post Last Implant | 3.04 (2.125) | 1.80 (1.792)
  6 Month Post Last Implant: number analyzed (Participants) | 8 | 8
  6 Month Post Last Implant | 4.96 (1.411) | 3.46 (1.040)

3. Secondary Outcome: Testosterone
Description: Long-term treatment with histrelin acetate suppresses the LH response to GnRH causing LH levels to decrease to prepubertal levels within 1 month of treatment. As a result, serum concentrations of sex steroids (estrogen or testosterone) also decrease. Testosterone suppression is defined as serum testosterone < 30.0 ng/dL (0.8 nmol/L) in boys following the induction of suppression. One black female participant age 8.9 years old had a testosterone value of 11ng/dL at visit 4 (month 6).
Time Frame: Baseline - 12 Months Post Last Implant
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: NG/DL
Arm/Group | Observed Value | Change From Baseline
Number analyzed (Participants) | 3 | 2
NG/DL
  Baseline: number analyzed (Participants) | 2 | 0
  Baseline | 10.95 (1.485) |
  Month 1, Visit 2: number analyzed (Participants) | 2 | 2
  Month 1, Visit 2 | 6.50 (2.687) | -4.45 (1.202)
  Month 3, Visit 3: number analyzed (Participants) | 2 | 2
  Month 3, Visit 3 | 8.25 (2.475) | -2.70 (0.990)
  Month 6, Visit 4 | 12.67 (2.082) | 2.55 (3.606)
  Month 9, Visit 5: number analyzed (Participants) | 2 | 2
  Month 9, Visit 5 | 8.15 (2.616) | -2.80 (1.131)
  Month 12, Visit 6: number analyzed (Participants) | 2 | 2
  Month 12, Visit 6 | 8.00 (4.243) | -2.95 (2.758)
  Month 13, Visit 7: number analyzed (Participants) | 1 | 1
  Month 13, Visit 7 | 14.00 | 2.00
  Month 18, Visit 9: number analyzed (Participants) | 2 | 2
  Month 18, Visit 9 | 9.80 (0.000) | -1.15 (1.485)
  Month 24, Visit 11: number analyzed (Participants) | 2 | 2
  Month 24, Visit 11 | 9.90 (4.384) | -1.05 (2.899)
  Month 36, Visit 13: number analyzed (Participants) | 1 | 1
  Month 36, Visit 13 | 6.90 | -3.00
  Month 42, Visit 14: number analyzed (Participants) | 1 | 1
  Month 42, Visit 14 | 8.10 | -1.80
  Month 48, Visit 15: number analyzed (Participants) | 1 | 1
  Month 48, Visit 15 | 7.30 | -2.60
  Month 54, Visit 16: number analyzed (Participants) | 1 | 1
  Month 54, Visit 16 | 4.10 | -5.80
  Month 60, Visit 17: number analyzed (Participants) | 1 | 1
  Month 60, Visit 17 | 7.00 | -2.90
  6 Months Post Last Implant: number analyzed (Participants) | 1 | 1
  6 Months Post Last Implant | 17.00 | 7.10
  12 Months Post Last Implant: number analyzed (Participants) | 1 | 1
  12 Months Post Last Implant | 130.00 | 120.10

4. Secondary Outcome: DHEA Sulfate
Description: DHEA=Dehydroepiandrosterone
Time Frame: Baseline - 36 Months Post Last Implant
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: UG/DL
Arm/Group | Observed Value | Change From Baseline
Number analyzed (Participants) | 31 | 31
UG/DL
  Baseline: number analyzed (Participants) | 26 | 0
  Baseline | 61.69 (36.526) |
  Month 3, Visit 3: number analyzed (Participants) | 16 | 15
  Month 3, Visit 3 | 70.88 (46.802) | 11.67 (15.281)
  Month 6, Visit 4: number analyzed (Participants) | 26 | 24
  Month 6, Visit 4 | 66.92 (36.739) | 6.08 (14.961)
  Month 9, Visit 5: number analyzed (Participants) | 27 | 25
  Month 9, Visit 5 | 71.22 (45.057) | 12.16 (15.085)
  Month 12, Visit 6: number analyzed (Participants) | 29 | 26
  Month 12, Visit 6 | 80.34 (48.207) | 25.77 (28.256)
  Month 13, Visit 7: number analyzed (Participants) | 27 | 24
  Month 13, Visit 7 | 81.00 (43.624) | 23.42 (23.178)
  Month 18, Visit 9: number analyzed (Participants) | 28 | 24
  Month 18, Visit 9 | 83.25 (47.973) | 27.79 (20.381)
  Month 24, Visit 11: number analyzed (Participants) | 29 | 26
  Month 24, Visit 11 | 87.31 (47.283) | 32.08 (34.599)
  Month 36, Visit 13: number analyzed (Participants) | 14 | 11
  Month 36, Visit 13 | 78.50 (72.809) | 37.45 (50.794)
  Month 42, Visit 14: number analyzed (Participants) | 10 | 7
  Month 42, Visit 14 | 49.00 (39.443) | 14.00 (28.537)
  Month 48, Visit 15: number analyzed (Participants) | 12 | 9
  Month 48, Visit 15 | 80.00 (50.292) | 36.56 (39.313)
  Month 54, Visit 16: number analyzed (Participants) | 5 | 3
  Month 54, Visit 16 | 60.60 (43.952) | 31.67 (22.723)
  Month 60, Visit 17: number analyzed (Participants) | 9 | 7
  Month 60, Visit 17 | 89.44 (34.667) | 53.14 (25.635)
  Month 66, Visit 18: number analyzed (Participants) | 2 | 1
  Month 66, Visit 18 | 57.50 (3.536) | 40.00
  Month 72, Visit 19: number analyzed (Participants) | 2 | 1
  Month 72, Visit 19 | 41.00 (4.243) | 23.00
  6 Months Post Last Implant: number analyzed (Participants) | 8 | 7
  6 Months Post Last Implant | 114.25 (50.692) | 61.43 (28.148)
  12 Months Post Last Implant: number analyzed (Participants) | 8 | 8
  12 Months Post Last Implant | 131.88 (69.907) | 71.00 (53.492)
  24 Months Post Last Implant: number analyzed (Participants) | 2 | 2
  24 Months Post Last Implant | 195.00 (98.995) | 140.50 (84.146)
  36 Months Post Last Implant: number analyzed (Participants) | 1 | 1
  36 Months Post Last Implant | 184.00 | 119.00

5. Secondary Outcome: Estradiol (MS)
Description: Long-term treatment with histrelin acetate suppresses the LH response to GnRH causing LH levels to decrease to prepubertal levels within 1 month of treatment. As a result, serum concentrations of sex steroids (estrogen or testosterone) also decrease. Estradiol suppression is defined as serum estradiol in the assay specific range < 20 pg/mL (73 pmol/L) in girls following the induction of suppression.
Time Frame: Month 36 - 36 Months Post Last Implant
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: NG/DL
Arm/Group | Observed Value
Number analyzed (Participants) | 12
NG/DL
  Month 36, Visit 13 | 0.46 (0.277)
  Month 42, Visit 14: number analyzed (Participants) | 9
  Month 42, Visit 14 | 0.38 (0.307)
  Month 48, Visit 15: number analyzed (Participants) | 11
  Month 48, Visit 15 | 0.52 (0.319)
  Month 54, Visit 16: number analyzed (Participants) | 4
  Month 54, Visit 16 | 0.47 (0.289)
  Month 60, Visit 17: number analyzed (Participants) | 7
  Month 60, Visit 17 | 0.50 (0.201)
  Month 66, Visit 18: number analyzed (Participants) | 2
  Month 66, Visit 18 | 0.21 (0.106)
  Month 72, Visit 19: number analyzed (Participants) | 2
  Month 72, Visit 19 | 0.34 (0.205)
  6 Months Post Last Implant: number analyzed (Participants) | 7
  6 Months Post Last Implant | 2.38 (0.909)
  12 Months Post Last Implant: number analyzed (Participants) | 7
  12 Months Post Last Implant | 4.00 (2.810)
  24 Months Post Last Implant: number analyzed (Participants) | 2
  24 Months Post Last Implant | 2.70 (0.424)
  36 Months Post Last Implant: number analyzed (Participants) | 1
  36 Months Post Last Implant | 3.10

6. Secondary Outcome: Estradiol (RIA)
Description: as for outcome 5
Time Frame: Baseline - Month 24
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: NG/DL
Arm/Group | Observed Value | Change From Baseline
Number analyzed (Participants) | 29 | 29
NG/DL
  Baseline: number analyzed (Participants) | 28 | 0
  Baseline | 1.58 (1.754) |
  Day 1, Visit 1: number analyzed (Participants) | 1 | 1
  Day 1, Visit 1 | 0.50 | 0.00
  Month 1, Visit 2: number analyzed (Participants) | 29 | 28
  Month 1, Visit 2 | 0.58 (0.199) | -1.00 (1.775)
  Month 3, Visit 3: number analyzed (Participants) | 29 | 28
  Month 3, Visit 3 | 0.55 (0.160) | -1.03 (1.765)
  Month 6, Visit 4: number analyzed (Participants) | 28 | 27
  Month 6, Visit 4 | 0.52 (0.061) | -1.10 (1.742)
  Month 9, Visit 5: number analyzed (Participants) | 28 | 27
  Month 9, Visit 5 | 0.55 (0.114) | -1.06 (1.794)
  Month 12, Visit 6: number analyzed (Participants) | 20 | 19
  Month 12, Visit 6 | 0.72 (0.526) | -0.62 (1.599)
  Month 13, Visit 7: number analyzed (Participants) | 27 | 27
  Month 13, Visit 7 | 0.57 (0.184) | -1.05 (1.806)
  Month 18, Visit 9: number analyzed (Participants) | 9 | 9
  Month 18, Visit 9 | 0.61 (0.154) | -0.69 (1.670)
  Month 24, Visit 11: number analyzed (Participants) | 9 | 9
  Month 24, Visit 11 | 0.61 (0.136) | -0.48 (1.119)

7. Secondary Outcome: Average Number of Implants Received
Description: There were 2 implants received that were not removed during the study and were excluded from this analysis due to unknown duration of treatment.
Time Frame: 12 months
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: Implants
Arm/Group | Histrelin Subcutaneous Implant (50 mg)
Number analyzed (Participants) | 31
Implants | 3.5 (1.36)

8. Secondary Outcome: Average Mean Implant Duration by Subject
Description: as for outcome 7
Time Frame: 12 Months
Population: Extension Safety Population
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Histrelin Subcutaneous Implant (50 mg)
Number analyzed (Participants) | 31
Months | 12.62 (0.469)

9. Secondary Outcome: Summary of EN3326 Implantation and Explantations
Description: Once the female participants reached 11 years of age and the male participants reached 12 years of age or the investigator determined that subjects no longer required hormone suppression, participants underwent final explantation and were eligible to continue into an optional Long Term Follow Up Phase (Post Implant Treatment Phase) for up to 5 years. The purpose of the optional Long Term Follow Up Phase was to collect additional medical and developmental information, such as onset of menses and final adult height after hormone suppression was discontinued.
Time Frame: Day 1 - Month 60
Population: Extension Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted | Removed
Number analyzed (Participants) | 31 | 31
Participants
  First Implant (Day 1, Visit 1) | 31 | 31
  Second Implant (Month 12, Visit 6) | 31 | 31
  Third Implant (Month 24, Visit 11) | 22 | 22
  Fourth Implant (Month 36, Visit 13) | 13 | 13
  Fifth Implant (Month 48, Visit 15) | 11 | 9
  Sixth Implant (Month 60, Visit 17) | 2 | 2

ADVERSE EVENTS:
Time Frame: From start of 2nd implant period through end of 6th implant period up to 48 months.
Arm/Group | Overall - Histrelin Subcutaneous Implant (50 mg)
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall - Histrelin Subcutaneous Implant (50 mg) (N=31)
Aggression (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall - Histrelin Subcutaneous Implant (50 mg) (N=31)
Implant Site Reaction (General disorders) | 20
Upper Respiratory Tract Infection (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 6
Pharyngitis Streptococcal (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Headache (Nervous system disorders) | 6
Weight Increased (Investigations) | 4
Agression (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No